CLINICAL TRIAL: NCT00810238
Title: C-Cure - Safety, Feasibility and Efficacy of Guided Bone Marrow-derived Mesenchymal Cardiopoietic Cells for the Treatment of Heart Failure Secondary to Ischemic Cardiomyopathy
Brief Title: C-Cure Clinical Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Celyad Oncology SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C3BS-C-07-01; EudraCT 2007-007699-40
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Heart Failure Class II or III
Keywords: Heart failure; Cell therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Optimal standard of care + C-Cure
  Interventions: Biological: C-Cure
- 2 (No Intervention): Optimal standard of care

INTERVENTIONS:
Biological: C-Cure — Intraventricular injection
  Arms: 1

SUMMARY:
The purpose of this clinical trial is to evaluate the feasibility, safety and efficacy of left ventricular endocardial injection of guided bone marrow-derived cardiopoietic cells (C-Cure) in the setting of chronic heart failure secondary to ischemic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 and < 75 years old;
* Subject has Heart Failure, New York Heart Association (NYHA) class II or class III with LVEF > 15% and ≤ 40% as assessed by transthoracic echocardiography;
* Subject has ischemic heart disease;
* Subject has an identifiable (by transthoracic echocardiography) area of transmural scar within the left ventricle;
* Subject is on optimal and stable medical therapy for more than 2 months;
* Subject is willing and able to undergo an ICD implantation, prior to receiving C-Cure™ or already has an ICD implanted;
* Subject agrees to comply with all follow-up evaluations;
* Subject has been informed of the nature of the clinical trial and agrees to its provision and has provided written informed consent.

Exclusion Criteria:

* Subject has been treated with cell-based therapy;
* Subject has myocardial revascularization by PCI or CABG within 2 months prior to enrolment;
* Subject has had an MI within 2 months prior to enrolment;
* Subject is planned for PCI, CABG or any cardiac surgery;
* Subject has received a biventricular pacemaker within 6 month prior to enrolment;
* Subject has moderate to severe aortic valve heart disease, aortic or mitral prosthetic valve;
* Subject has a significant mitral valve insufficiency (Effective Regurgitant Orifice (ERO) > 0.2 cm²) with possibility of mitral valve surgery;
* Subject has left ventricular thrombus;
* Subject has LV aneurysma or is a candidate for surgical aneurysmectomy;
* Subject LV ventricular wall thickness is < 5 mm in the target territory;
* Subject has proven high grade atrioventricular block or sustained ventricular tachyarrhythmias;
* Subject has an hemodynamically significant congenital heart disorder;
* Subject has clinical evidence for infection or active malignancy;
* Subject has known stable chronic kidney dysfunction with serum creatinine > 2.5 mg/dL at two occasions during the screening period;
* Subject has experienced severe adverse reaction/allergies to contrast agents;
* Subject has atherosclerosis and/or tortuosity of the aorta, iliac or femoral arteries of a degree, that could impede or preclude the safe retrograde passage of the delivery catheter, in the judgment of the investigator;
* Subject is on chronic immunosuppressive transplant therapy;
* Subject had an autologous or allogenic bone marrow or peripheral stem cell transplant or prior solid organ transplantation;
* Subject has a multisystem disease;
* Subject has been tested positive for Human Immunodeficiency Virus (HIV 1 or HIV 2), Hepatitis B Virus (HBV), Hepatitis C (HCV) and/or syphilis;
* Women of child bearing potential;
* Subject has life expectancy < 1 year from non heart failure related causes;
* Subject suffers from morbid obesity (Body Mass Index (BMI) > 40);
* Subject has a recent history of alcohol or drug abuse;
* Subject has any other surgical or medical condition that, in the judgment of the investigator might warrant exclusion or be contraindicated for safety reasons;
* Subject is currently participating in another trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction | 6 months

SECONDARY OUTCOMES:
6-min walking distance | 6 months, 1 and 2 years
Quality of Life | 6 months, 1 and 2 years
All cause mortality | Each follow-up
Cardiovascular events | Each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Bartunek, MD, PhD, Principal Investigator — VZW Cardiovascular Research Center Aalst; André Terzic, MD, PhD, Principal Investigator — Mayo Clinic, Rochester, USA
Locations (8):
- Belgium (7):
  - CardioVascular Center, Aalst
  - Université Catholique de Louvain, Saint-Luc, Brussels
  - Centre Hospitalier Universitaire, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ziekenhuis Oost Limburg, Genk
  - Virga Jesse Ziekenhuis, Hasselt
  - Centre Hospitalier Universitaire, Liège
- Clinical Center of Serbia, Belgrade, Serbia

REFERENCES:
- [Derived] Bartunek J, Behfar A, Dolatabadi D, Vanderheyden M, Ostojic M, Dens J, El Nakadi B, Banovic M, Beleslin B, Vrolix M, Legrand V, Vrints C, Vanoverschelde JL, Crespo-Diaz R, Homsy C, Tendera M, Waldman S, Wijns W, Terzic A. Cardiopoietic stem cell therapy in heart failure: the C-CURE (Cardiopoietic stem Cell therapy in heart failURE) multicenter randomized trial with lineage-specified biologics. J Am Coll Cardiol. 2013 Jun 11;61(23):2329-38. doi: 10.1016/j.jacc.2013.02.071. Epub 2013 Apr 10. PMID 23583246